CLINICAL TRIAL: NCT06469437
Title: The Impact of Geriatric Assessment on the Treatment Plan of Elderly Patients With Type 2 Diabetes Mellitus: a Randomized Clinical Trial.
Brief Title: The Impact of Geriatric Assessment on the Treatment Plan of Elderly Patients With T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0456
Record Dates: First submitted 2024-05-13; First posted 2024-06-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Type2diabetes; Frail Elderly Syndrome; Frailty; Geriatric Assessment
Keywords: Type 2 diabetes; Frailty; Geriatric assessement; Glycated hemoglobin
MeSH Terms: conditions — Frailty; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This group will be submitted to geriatric assessment through CFS and TaGA-10 tools only.
- Intervention (Experimental): This group will be submitted to geriatric assessment through CFS and TaGA-10 tools, and the investigators will provide the physician with a short note with the proposed glycated hemoglobin target.
  Interventions: Behavioral: Providing the physicians with a proposed glycated hemoglobin target

INTERVENTIONS:
Behavioral: Providing the physicians with a proposed glycated hemoglobin target — Through the geriatric assessment, the investigators will categorize the groups proposed by the Diabetes Canada Clinical Practice Guidelines Expert Committee guideline recommendations into "functionally independent", "functionally dependent" and "frail". The investigators will provide the physician with the glycated hemoglobin target proposed by the guideline.
  Arms: Intervention

SUMMARY:
Introduction: With the aging of the world population and the increasing incidence of type 2 diabetes mellitus (T2DM) with age, the number of elderly individuals living with diabetes has been considerably rising. It is known that uncontrolled T2DM negatively impacts various health outcomes, including geriatric outcomes such as sarcopenia, frailty, immobility, incontinence, and infections. Current medical literature fails to establish appropriate glycemic targets for different elderly profiles. Although guidelines emphasize the need to individualize targets, there is no concise tool to identify which individuals benefit from each therapeutic approach. Data suggest that frailty is the best predictor of negative outcomes in elderly patients living with T2DM. The Clinical Frailty Scale (CFS) and the 10-minute Targeted Geriatric Assessment (TaGA-10) are validated tools for prognosis in elderly patients and for identifying frail elderly individuals.

Methods: Randomized controlled trial. Elderly individuals diagnosed with T2DM at a tertiary care outpatient clinic will be included. All enrolled patients will undergo geriatric assessment using CFS, TaGA-10, and Charlson Comorbidity Index. Patients will be randomized into usual care and intervention groups, and the intervention involves providing the geriatric assessment to the care team to support their decisions. The adequacy of the therapeutic approach will be measured in one week by reviewing the consult record or interviewing the physician. The clinical impact on the frequency of hypoglycemia, falls, infections, hospitalizations, and mortality will be evaluated at 3 and 6 months by telephone interviews.

Discussion: Current guidelines recommend using age, comorbidities, cognitive, and functional status to individualize therapeutic targets in elderly patients with T2DM; however, it is possible that these variables alone may not be sufficient to classify all elderly individuals in their complexity adequately. A tool with such power and easy to use in clinical practice is necessary.

DETAILED DESCRIPTION:
All patients included in the research (both intervention and control groups, totaling a sample size of N=220 participants) will undergo geriatric assessment using the CFS and TaGA-10 tools. Using the CFS, the investigators will classify patients with scores of 1 to 3 as "functionally independent," 4 to 5 as "functionally dependent," and scores 6 to 8 as "frail." Patients will be randomized by random permuted block randomization, with block sizes of 2 and 4, stratified by frailty status ("functionally independent", "functionally dependent", or "frail").

Patients allocated to the control group will receive usual treatment without any additional procedures.

For the intervention group, before making decisions in the case discussion, the investigators will provide the physician a short note containing a suggested care plan as follows:

* Functionally independent (CFS 1-3): Glycemic targets should be equal to the general population, disregarding age. Consider seeking long-term treatment effects. Target suggested HbA1c around 7.0%.
* Functionally dependent (CFS 4-5): Consider higher glycemic targets by 0.5% compared to the general adult population. Aim for short- and medium-term treatment effects. Target suggested HbA1c less than 8.0%.
* Frail (CFS 6-8): Consider higher glycemic targets by 1.5% compared to the general adult population. Aim to reduce treatment complications. Do not expect medium- and long-term treatment effects. Target suggested HbA1c less than 8.5%.

These care plans are based on the Diabetes Canada Clinical Practice Guidelines Expert Committee guideline recommendations. Patients with a CFS of 9 will be excluded due to the recommendation of not measuring HbA1c to this group.

The investigators will initially approach the physicians at the outpatient clinic to apply the informed consent process and request possible eligible patients from the physician. Each physician will sign a consent form to participate in the entire study. Afterward, the investigators will check the patient's eligibility and apply the informed consent. If any of the participants (physician or patient) disagree with participating in the research, the pair will not be included. Physicians and patients wishing to withdraw consent to participate in the research can do so at any time; in this case, the pair will be treated as lost to follow-up.

The application of the Clinical Frailty Scale, with an estimated duration of 1 minute, will be conducted immediately after obtaining informed consent from the patient. The physician will attend to the patient, and during the discussion with the preceptor, the investigators will apply the TaGA-10 scale in the office. At this time, the patient will also be randomized with the assistance of the RedCap program. For the intervention group, the investigators will provide the physician with a geriatric assessment proposing a glycated hemoglobin target.

Information not requiring in-person assessment will be collected from medical records or during a telephone interview. The adequacy of the therapeutic approach (main outcome) will be measured in one week by reviewing the consult record or interviewing the physician.

The second and third evaluations will be conducted by telephone contact 3 and 6 months after the first visit. During this contact, the incidence of falls, infections, hypoglycemia, hospitalizations, and death will be queried, as long as the consult of new measurements of HbA1c on medical records. The data will be stored using the institutional computer in the institutional Google Drive and will be processed and analyzed using the RedCap program. The data will be anonymized for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Diagnostic of type 2 diabetes mellitus according to American Diabetes Association criteria
* Patients under follow-up in a specialized endocrinology outpatient clinic
* Patients who have a glycated hemoglobin measurement of up to one month

Exclusion Criteria:

* Lack of consent for research participation from the patient or the physician
* Patients classified as Clinical Frailty Scale 9.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adequacy of hyperglycemia prescription | up to 1 week
  The adequacy of treatment will be considered when:
  * The treatment is intensified if the patient's HbA1C is higher by at least 0.5% than the glycemic target proposed by the geriatric assessment.
  * The treatment is de-intensified if the patient's HbA1C is lower by at least 0.5% than the glycemic target proposed by the geriatric assessment.
  * The treatment is maintained if the patient's HbA1C is within 0.5% above or below the glycemic target proposed by the geriatric assessment.

SECONDARY OUTCOMES:
Hypoglycemia (general and severe) | up to 6 months.
  Hypoglycemia is defined by blood sugar levels below 70mg/dl and severe hypoglycemia requires assistance from another person. This outcome will be assessed through a questionnaire administered to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Incidence of falls | up to 6 months.
  Number of falls in general and the number of falls that require emergency care. This outcome will be assessed through a questionnaire administered to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Infection | up to 6 months.
  Number of infections requiring antibiotics prescription. Severe infection will be considered when hospitalization is needed. This outcome will be assessed through a questionnaire administered to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Hospitalization | up to 6 months.
  Number of times the patient required hospitalization in general and due to diabetes. This outcome will be assessed through a questionnaire administered to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Death | up to 6 months.
  This outcome will be assessed through a questionnaire to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Adequacy of antiplatelet prescription | up to 6 months.
  Based on medical records, the investigators will measure the adequacy of antiplatelet prescription. This outcome will be assessed through a questionnaire administered to the patient or family member in a telephone interview one month after the second consultation (approximately 6 months after the index consultation).
Glycemic control | up to 6 months.
  Based on medical records, the investigators will consult if the patient have new measurements of glycated hemoglobin and its adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Renato GB Mello, Professor, Principal Investigator — Federal University of Rio Grande do Sul; Dimitris RV Rados, Professor, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sesti G, Antonelli Incalzi R, Bonora E, Consoli A, Giaccari A, Maggi S, Paolisso G, Purrello F, Vendemiale G, Ferrara N. Management of diabetes in older adults. Nutr Metab Cardiovasc Dis. 2018 Mar;28(3):206-218. doi: 10.1016/j.numecd.2017.11.007. Epub 2017 Dec 7. PMID 29337017
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Strain WD, Hope SV, Green A, Kar P, Valabhji J, Sinclair AJ. Type 2 diabetes mellitus in older people: a brief statement of key principles of modern day management including the assessment of frailty. A national collaborative stakeholder initiative. Diabet Med. 2018 Jul;35(7):838-845. doi: 10.1111/dme.13644. Epub 2018 May 6. PMID 29633351
- [Background] Hubbard RE, Andrew MK, Fallah N, Rockwood K. Comparison of the prognostic importance of diagnosed diabetes, co-morbidity and frailty in older people. Diabet Med. 2010 May;27(5):603-6. doi: 10.1111/j.1464-5491.2010.02977.x. PMID 20536960
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Meneilly GS, Knip A, Miller DB, Sherifali D, Tessier D, Zahedi A. Diabetes in Older People. Can J Diabetes. 2018 Apr;42 Suppl 1:S283-S295. doi: 10.1016/j.jcjd.2017.10.021. No abstract available. PMID 29650107
- [Background] MacKenzie HT, Tugwell B, Rockwood K, Theou O. Frailty and Diabetes in Older Hospitalized Adults: The Case for Routine Frailty Assessment. Can J Diabetes. 2020 Apr;44(3):241-245.e1. doi: 10.1016/j.jcjd.2019.07.001. Epub 2019 Jul 6. PMID 31466827
- [Background] Aliberti MJR, Covinsky KE, Apolinario D, Lee SJ, Fortes-Filho SQ, Melo JA, Viana SSC, Suemoto CK, Jacob-Filho W. A 10-min Targeted Geriatric Assessment Predicts Mortality in Fast-Paced Acute Care Settings: A Prospective Cohort Study. J Nutr Health Aging. 2019;23(3):286-290. doi: 10.1007/s12603-018-1152-z. PMID 30820518